CLINICAL TRIAL: NCT00363805
Title: Chemoprevention of Lung Carcinogenesis Using Green Tea: Phase IIb Randomized, Double-Blinded, Placebo Controlled Trial of Green Tea and Polyphenon E in Former Smokers With Chronic Obstructive Lung Disease (COPD)
Brief Title: Green Tea or Polyphenon E in Preventing Lung Cancer in Former Smokers With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sherry Chow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sherry Chow, Research Professor, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDR0000487501; U01CA101204 (NIH); P30CA023074 (NIH); UARIZ-HSC-0353
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Lung Cancer Prevention
Keywords: lung cancer; prevention; green tea; former smokers
MeSH Terms: conditions — Lung Neoplasms; Smoking Cessation | interventions — Tea; polyphenon E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Green Tea (Experimental): Patients receive green tea beverage and placebo capsules for 6 months.
  Interventions: Dietary Supplement: green tea
- Polyphenon E (Experimental): Patients receive placebo beverage and Polyphenon E capsules daily for 6 months.
  Interventions: Drug: Polyphenon E
- Placebo (Placebo Comparator): Patients receive placebo beverage and placebo capsules daily for 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: green tea — Given orally
  Arms: Green Tea
Drug: Polyphenon E — Given orally
  Arms: Polyphenon E
Other: placebo — Given orally
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention is the use of certain substances to keep cancer from forming, growing, or coming back. The use of green tea or polyphenon E may prevent cancer from forming in former smokers with chronic obstructive pulmonary disease.

PURPOSE: This randomized phase II trial is studying how well green tea or polyphenon E work in preventing lung cancer in former smokers with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effects of high-level oral consumption of defined green tea (four 12-oz servings/day) or polyphenon E capsules (4 capsules/day) on markers of cellular oxidative damage, as measured by 8-hydroxydeoxyguanosine (8-OHdG) and 8-F_2-isoprostanes (8-epi-PGF2) in former smokers with chronic obstructive pulmonary disease.

Secondary

* Evaluate the effects of high-level oral consumption of defined green tea or polyphenon E capsules on body antioxidant status (carotenoids, vitamins A and E, ascorbic acid [vitamin C] and antioxidant enzymes [catalase and glutathione peroxidase]) in blood in these patients.
* Evaluate the effects of high-level oral consumption of defined green tea or polyphenon E capsules on gene expression of markers of proliferation and apoptosis in induced sputum in these patients.

Tertiary

* Evaluate the effects of high-level oral consumption of defined green tea or polyphenon E capsules on lung function in these patients.
* Evaluate the relative adherence to use of green tea beverage vs polyphenon E capsules in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to gender and inhaled steroid usage (yes vs no).

All patients receive placebo tea beverage and placebo capsules 4 times a day for 2 weeks. Patients are randomized to 1 of 3 treatment arms after successful completion of the 2-week period.

* Arm I (green tea beverage): Patients receive oral green tea beverage and oral polyphenon E placebo daily for 6 months.
* Arm II (green tea capsule [polyphenon E]): Patients receive oral green tea beverage placebo and oral polyphenon E daily for 6 months.
* Arm III (placebo): Patients receive oral green tea beverage placebo and oral polyphenon E placebo daily for 6 months.

Patients undergo blood, urine, exhaled breath condensate (EBC), induced sputum, and buccal cell collection at baseline and periodically during study for biomarker/laboratory analysis. Blood samples are analyzed for 8-hydroxydeoxyguanosine (8-OHdG), glutathione peroxidase, and catalase. Urine is examined for F_2-isoprostanes, 8-OHdG, and tea polyphenols. Induced sputum broncho-epithelial cells are analyzed for gene expression of genes implicated in cellular growth and apoptotic pathway via reverse transcriptase-polymerase chain reaction. EBC samples are examined for F_2-isoprostane levels. Buccal cells are stored for future analysis.

PROJECTED ACCRUAL: A total of 195 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic obstructive pulmonary disease

  * FEV_1/FVC ≤ 78
* History of smoking ≥ 1 pack daily for 30 years OR 2 packs daily for 15 years

  * Stopped smoking for ≥ 1 year
* No previously diagnosed bronchiectasis
* No history of > 1 acute emphysema exacerbation within the past 3 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,500/mm³
* Platelet count > 130,000/mm³
* Hemoglobin ≥ 11 g/dL (female) or 12 g/dL (male)
* AST and ALT normal
* Bilirubin ≤ 1.5 mg/dL (unless Gilbert's disease present)
* Creatinine ≤ 1.5 mg/dL
* Alkaline phosphatase ≤ 2 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No invasive cancer within the past 5 years
* Able and willing to consume caffeinated beverages
* Able to produce induced sputum
* Able to perform forced expiratory maneuver during spirometry testing
* No immunosuppression by virtue of medication or disease including, but no limited to, any of the following:

  * Organ transplantation
  * Liver or kidney failure
  * Autoimmune diseases
  * Oral steroids
  * Chemotherapy
* No serious concurrent illness that could preclude study compliance, such as uncontrolled high blood pressure, heart disease, or poorly controlled diabetes
* No myocardial infarction within the past 6 weeks

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior and no concurrent dietary supplements or herbal products, including any of the following:

  * Herbal tea
  * Ginkgo biloba > 60 mg/day
  * Melatonin > 3 mg/day
  * Echinacea > 300 mg/day
  * Hypericum perforatum (St. John's wort) > 300 mg/day
  * DHEA mustard > 5 mg/day
* At least 2 weeks since prior and no concurrent nontrial tea or tea products
* More than 3 weeks since prior chest or abdominal surgery
* More than 3 months since prior participation in chemoprevention or clinical intervention trials
* At least 3 months since prior and no concurrent megadoses of vitamins, defined as > 4,000 IU of vitamin A, 400 IU of vitamin E, 400 IU of cholecalciferol (vitamin D), 60 μg of selenium, or 1,000 mg of ascorbic acid (vitamin C) per day
* No regular consumption of ≥ 6 cups or glasses of tea per week
* No concurrent nontrial caffeine at > 1 serving/day (1 serving defined as 12 oz of regular soda or 8 oz of coffee)
* No concurrent participation in another interventional clinical trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2004-05; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iman Hakim, MD, PhD, MPH, Principal Investigator — University of Arizona
Locations (3):
- United States (3):
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Tucson, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Green Tea | Polyphenon E | Placebo
Started | 42 | 63 | 73
Completed | 38 | 57 | 70
Not Completed | 4 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Green Tea | Polyphenon E | Placebo | Total
Number analyzed (Participants) | 42 | 63 | 73 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 34 | 35 | 85
  >=65 years | 26 | 29 | 38 | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.2) | 63.6 (8.5) | 64.3 (7.8) | 64.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 31 | 37 | 89
  Male | 21 | 32 | 36 | 89
Region of Enrollment [Number; unit: participants]
  United States | 42 | 63 | 73 | 178

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary 8-hydroxydeoxyguanosine Levels
Description: the urinary concentrations of 8-hydroxydeoxyguanosine were normalized by the urinary creatinine concentrations to correct for variations in urine dilution/production and the change in urinary 8-hydroxydeoxyguanosine levels was calculated as the 6 months levels minus the baseline levels
Time Frame: Baseline and 6 months
Population: The number of participants analyzed was less than the number of participants completing the study because the analysis only included samples where the identify of the analyte was confirmed in the sample.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Green Tea | Polyphenon E | Placebo
Number analyzed (Participants) | 33 | 51 | 67
ng/mg creatinine | 2.36 (10.48) | 5.20 (36.20) | -1.08 (25.41)

2. Primary Outcome: Change in Urinary 8-F2-isoprostanes Levels
Description: the urinary concentrations of 8-F2-isoprostanes were normalized by the urinary creatinine concentrations to correct for variations in urine dilution/production and the change in urinary 8-F2-isoprostanes levels was calculated as 6 months levels minus baseline levels
Time Frame: Baseline and 6 months
Population: The number of participants analyzed was less than the number of participants completing the study because the analysis only included samples where the identity of the analyte was confirmed in the sample.
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Green Tea | Polyphenon E | Placebo
Number analyzed (Participants) | 30 | 51 | 66
ng/mg creatinine | -39.87 (271.2) | -35.80 (261.7) | 0.71 (266.4)

ADVERSE EVENTS:
Arm/Group | Green Tea | Polyphenon E | Placebo
Serious Adverse Events (participants affected / at risk) | 4/42 | 4/63 | 7/73
Other Adverse Events (participants affected / at risk) | 12/42 | 14/63 | 21/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Green Tea (N=42) | Polyphenon E (N=63) | Placebo (N=73)
cardiac arrest (Cardiac disorders) | 0 | 0 | 1
chest pain (Cardiac disorders) | 0 | 0 | 1
other - knee surgery (Surgical and medical procedures) | 0 | 0 | 1
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
other - emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
bronchial infection (Infections and infestations) | 1 | 1 | 0
other - pneumonia (Infections and infestations) | 0 | 0 | 1
Flu-like symptoms (General disorders) | 1 | 0 | 0
pacemaker placement (Cardiac disorders) | 1 | 0 | 0
Other - replacement of implant stimulator in abdomen (Surgical and medical procedures) | 0 | 0 | 1
Other - surgery for unclogging carotid artery (Surgical and medical procedures) | 0 | 0 | 1
Other - knee replacement (Surgical and medical procedures) | 1 | 0 | 0
Other - placement of coronary stent (Surgical and medical procedures) | 0 | 1 | 0
Other - surgery on right ankle (Surgical and medical procedures) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Other - blood clotting disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Green Tea (N=42) | Polyphenon E (N=63) | Placebo (N=73)
dizziness (Nervous system disorders) | 4 | 2 | 3
headache (Nervous system disorders) | 4 | 4 | 4
Flu-like symptoms (General disorders) | 6 | 8 | 13
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3
dyspepsia (Gastrointestinal disorders) | 2 | 4 | 4
gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 3 | 1
nausea (Gastrointestinal disorders) | 4 | 3 | 0
constipation (Gastrointestinal disorders) | 0 | 4 | 0
hypertension (Vascular disorders) | 3 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No